CLINICAL TRIAL: NCT05880381
Title: Adaptive Virtual Reality for Coping With Involuntary Early Pregnancy Loss
Brief Title: Virtual Reality for Coping With Involuntary Early Pregnancy Loss
Acronym: AViR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Madeira (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Serviço de Saúde da Região Autónoma da Madeira- SESARAM (Unknown)
Responsible Party: Principal Investigator, Mónica Cameirão, Assistant Professor and researcher at the University of Madeira, Universidade da Madeira
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07/2023
Record Dates: First submitted 2023-04-17; First posted 2023-05-30 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Early Pregnancy Loss
Keywords: Virtual Reality; Psychological Intervention; Personalization
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of the two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Patients allocated to the treatment group will undergo an intervention that comprises 3 weekly sessions of 60 minutes for 4 weeks with the VR prototype.
  Interventions: Device: Virtual Reality Group
- Control Group (Other): The participants allocated to this group will do the formal standard care provided by the Gynecology- Obstetric service.
  Interventions: Other: Control Group

INTERVENTIONS:
Device: Virtual Reality Group — Patients allocated to the treatment group will undergo an intervention that comprises 3 weekly sessions of 60 minutes for 4 weeks with the VR prototype.
  Arms: Virtual Reality Group
Other: Control Group — The participants allocated to this group will do the formal standard care provided by the Gynecology- Obstetric service.
  Arms: Control Group

SUMMARY:
This study aims to provide psychological support to women that experienced an Early Pregnancy Loss (when the loss occurs until the 20 weeks of gestation) using an innovative Virtual Reality prototype and compare the presence and evolution of psychological distress symptoms pre and post-intervention.

The main goals of this study are:

1. Evaluate the impact of the proposed VR paradigm in women who suffered a gestational loss in the first 20 weeks of gestation, compared to a control group that follows the usual standard care;
2. Evaluate the usability, user experience, and acceptance of the proposed approach.

Participants in the VR group will have an intervention program lasting four weeks, with 3 weekly sessions of 45-60 minutes, using the developed prototype.

DETAILED DESCRIPTION:
Early pregnancy loss occurs in about 20% of all pregnancies and can lead to chronic grief and psychological distress symptomatology. Although the high prevalence, it is still a very undervalued event, and proper follow-up and psychological guidance are often absent.

The present research study aims to evaluate the feasibility of a psychological VR-based approach in a controlled pilot study with 20 women who suffered an early gestational loss in the last 6 months. Using the developed prototype, the experimental VR group will have an intervention program lasting four weeks, with 3 weekly sessions of 45-60 minutes.

The investigators aimed to verify if the use of the proposed VR paradigm will significantly reduce symptoms of grief, depression, anxiety and post-traumatic stress, and that this reduction will be significantly greater compared to the control group.

The study proposed is very innovative in terms of the target population and the use of VR, specifically designed to address gestational loss. In addition, it opens a new avenue of research on a topic that is still silenced and considered taboo in society. Thus, this interdisciplinary research has an expected scientific, technological, and social impact, namely: 1) contributes to a better understanding of the process of psychological recovery after an early gestational loss; 2) contributes to the advancement of technologies aimed at psychological support; 3) has the potential to accelerate the resolution of grief by bringing emotional and psychological support to women who do not have access to other means of support; and 4) contributes to reducing the economic burden on health care by providing tools to improve the well-being of patients.

ELIGIBILITY:
Inclusion Criteria:

- Women that have experienced an involuntary pregnancy loss in the first 20 weeks in the last 6 months;

Exclusion Criteria:

* current pregnancy
* having a diagnosis of mental disorder,
* undergoing any psychological intervention,
* vision impairments that could interfere with the execution of the VR tasks.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Perinatal Grief Scale (PGS) | Pre-intervention (1 week before the beginning of the intervention) and Post-intervention (4 to 5 weeks after the beginning of the intervention)
  Portuguese adaptation of Perinatal Grief Scale- PGS (Rocha, 2004) assesses changes pre and post-intervention, in three subscales that involve perinatal grief symptomatology like active grief, difficulty coping and despair. This scale comprises 33 items divided into three subscales that assess active grief, difficulty coping, and despair. Minimum score of 33 and a maximum 165- higher scores represent more severe grief symptoms.
Posttraumatic Stress Disorder Checklist (PCL-5) | Pre-intervention (1 week before the beginning of the intervention) and Post-intervention (4 to 5 weeks after the beginning of the intervention)
  The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5) adapted to the Portuguese population, will be used to evaluate post-intervention changes in post-traumatic stress symptoms. This is a 20-item self-report instrument that assesses the 20 DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) symptoms of PTSD rated from 0 to 4. A minimum score of 0 and a maximum of 80- higher scores represent more severe post-traumatic stress symptoms.
Hospital Anxiety and Depression Scale (HADS) | Pre-intervention (1 week before the beginning of the intervention) and Post-intervention (4 to 5 weeks after the beginning of the intervention)
  HADS is a 14-question instrument that measures anxiety and depression with seven questions for each; each question is scored between zero (no impairment) and three (severe impairment), with a maximum score of 21 for anxiety or depression.

SECONDARY OUTCOMES:
System Usability Scale (SUS) | Post-Intervention (4-5 weeks after the beginning of the intervention)
  For assessing the overall usability of the prototype, the System Usability Scale (SUS) is a widely used scale that provides a global view of subjective assessments of usability. Scoring varies from 0 to 100, and the bigger the value better the usability assessment.
Sense of Presence Inventory (ITC) | Post-Intervention (4-5 weeks after the beginning of the intervention)
  To assess the VR user experience, the ITC - Sense of Presence Inventory adapted to the Portuguese population by Raposo-Vasconcelos et al. will be used. This scale has two parts, the first addressing the user's feelings after the experience, and the second related to the characterization of the experience during the simulation. This inventory includes 44 items organized into four factors: Sense of physical space, Engagement, Ecological validity, and Negative effects. The mean score for each factor can vary from 1 to 5.
User Experience questionnaire | Post-Intervention (4-5 weeks after the beginning of the intervention)
  A customized questionnaire with open questions where participants can freely elaborate on any issues related to the VR prototype. Only qualitative data will be analysed with this questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade da Madeira, Funchal, Portugal

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT05880381/Prot_ICF_000.pdf